CLINICAL TRIAL: NCT02825355
Title: Sentinel Node Mapping With Robotic Assisted Near Infra-red Fluorescent Imaging in Women With Cervical and Endometrial Cancer
Brief Title: Sentinel Node Mapping in Women With Cervical and Endometrial Cancer
Acronym: SENTIREC I
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Sara Sponholtz, MD, University of Southern Denmark
Other Study IDs: SDUSF12015163 1 (198)
Record Dates: First submitted 2016-06-23; First posted 2016-07-07 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Uterine Cervical Neoplasms; Uterine Neoplasms
Keywords: robotic surgery procedure; indocyanine green; sentinel lymph node mapping
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with cervical cancer: All patients receive sentinel node mapping as the conventional treatment.
- Patients with endometrial cancer: All patients receive sentinel node mapping as the conventional treatment.

SUMMARY:
This study aims to evaluate the effect of SLN mapping on the incidence and severity of lymphedema in women with early stage cervical and endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Study IA: Cervical carcinoma, FIGO stage IB1, cervical tumour size < 2 cm
* Study IB: Endometrial adenocarcinoma, presumed FIGO stage I, low- and intermediate risk: Type 1 grade 1 + 2, > 50% myometrial invasion

Exclusion Criteria:

* Prior PL
* Known allergy towards ICG and/or iodine (ICG contains 5% sodium iodine)
* Women included in other studies affecting outcome-measures of the present study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See above in eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of lymphedema | 3 years
  Incidence of lymphedema will be assessed using patient reported outcome measures.
Severity of lymphedema | 3 years
  Severity of lymphedema will be assessed using patient reported outcome measures.

SECONDARY OUTCOMES:
Detection rate of sentinel lymph node | 2 years
  Detection of sentinel lymph node per patient, per heme-pelvis and bilaterally
Mapping of SLN in different types of lymph node stations | 2 years
  Mapping of SLN in areas outside the normal area of pelvic lymphadenectomy

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Bjornholt SM, Sponholtz SE, Markauskas A, Froding LP, Larsen CR, Fuglsang K, Schledermann D, Mogensen O, Jensen PT. Sentinel lymph node mapping for endometrial and cervical cancer in Denmark. Dan Med J. 2021 Mar 24;68(4):A11200886. PMID 33829991